CLINICAL TRIAL: NCT04973605
Title: A Phase 1b/2 Dose-Escalation and Cohort-Expansion Study to Determine the Safety and Efficacy of BGB-11417as Monotherapy, in Combination With Dexamethasone, Dexamethasone/Carfilzomib, Dexamethasone/Daratumumab, and Dexamethasone/Pomalidomide in Patients With Relapsed/Refractory Multiple Myeloma and t(11;14)
Brief Title: A Phase 1b/2 Study of Sonrotoclax (BGB-11417) as Monotherapy and in Various Combinations With Dexamethasone Plus Carfilzomib, Dexamethasone Plus Daratumumab, and Dexamethasone Plus Pomalidomide in Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417-105; 2023-507751-30-00 (EU CTIS Number); 2021-003614-39 (EudraCT Number); U1111-1277-5444 (Other: UTN Number); CTR20231932 (Other: ChinaDrugTrials)
Record Dates: First submitted 2021-07-07; First posted 2021-07-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-02

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; carfilzomib; daratumumab; pomalidomide

STUDY DESIGN:
Intervention Model Description: Participants will be assigned sequentially in Part 1. In Part 2 participants will be assigned in parallel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 Dose Escalation (Experimental): Dose-escalation and de-escalation to determine maximum tolerated dose (MTD) of sonrotoclax plus dexamethasone, sonrotoclax plus dexamethasone plus carfilzomib, sonrotoclax plus dexamethasone plus daratumumab, and sonrotoclax plus dexamethasone plus pomalidomide.
  Interventions: Drug: Sonrotoclax; Drug: Dexamethasone; Drug: Carfilzomib; Drug: Daratumumab; Drug: Pomalidomide
- Part 2 Cohort Expansion (Experimental): There will be up to 7 expansion cohorts to further evaluate the safety and efficacy of sonrotoclax monotherapy, sonrotoclax plus dexamethasone in combination with dexamethasone plus carfilzomib, and in combination with dexamethasone plus daratumumab
  Interventions: Drug: Sonrotoclax; Drug: Dexamethasone; Drug: Carfilzomib

INTERVENTIONS:
Drug: Sonrotoclax — Administered orally daily
  Other Names: BGB-11417
Drug: Dexamethasone — Once weekly either orally or intravenously
Drug: Carfilzomib — Administered intravenously weekly
Drug: Daratumumab — Administered subcutaneously weekly
  Arms: Part 1 Dose Escalation
Drug: Pomalidomide — Administered orally daily
  Arms: Part 1 Dose Escalation

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and efficacy of sonrotoclax as monotherapy and in various combinations in patients with relapsed/refractory (R/R) multiple myeloma (MM) and chromosomal translocation t(11;14).

The study investigates sonrotoclax alone and in combination with dexamethasone and other agents, including carfilzomib, daratumumab, and pomalidomide.

DETAILED DESCRIPTION:
Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
2. A confirmed diagnosis of multiple myeloma (must have an M-component in serum and/or urine)
3. Measurable disease defined as:

   i. M-spike ≥ 500mg/dL, or ii. Urine protein M-spike of ≥ 200 mg/day, or iii. Serum free light chains ≥ 10 mg/dL, and an abnormal κ:λ ratio
4. Participant has documented relapsed or progressive MM on or after any regimen or who are refractory to the most recent line of therapy.

   i. Relapsed MM is defined as previously treated MM that progresses and requires initiation of salvage therapy but does not meet the criteria for refractory MM.

   ii. Refractory MM is defined as disease that is nonresponsive (failure to achieve minimal response or development of progressive disease) while on primary or salvage therapy or progresses within 60 days of last therapy.
   1. In Part 1 and Part 2 Cohorts 1 and 2 participants should have relapsed or progressive disease and have had ≥ 3 prior lines of therapy including a proteasome inhibitor, an IMiD, and an anti-CD38 monoclonal antibody, and no more available approved therapies.
   2. Participants in Part 2 Cohorts 3, 4, and 5 should have relapsed or progressive disease and have had ≥ 1 prior line of therapy. Prior treatment with carfilzomib is allowed but the patient must not be considered carfilzomib refractory by the investigator.
   3. Participants in Part 2 Cohorts 6 and 7 should have relapsed or progressive disease and have had 1 to 3 prior lines of therapy and previously treated with a proteasome inhibitor and an IMiD
5. Positivity for t(11;14) translocation must be confirmed by validated fluorescence in situ hybridization (FISH) testing assay in a pre-defined laboratory

   a. fresh bone marrow aspirate sample must be collected at screening and sent to central laboratory for t(11;14) FISH testing.
6. Adequate organ function defined as:

   1. Hemoglobin ≥ 8.0 g/dL within 7 days before first dose of study treatment, (transfusions, in accordance with institutional guidelines, are permitted)
   2. Platelet count ≥ 75,000/μL, within 7 days before first dose of study treatment, independent of growth factor support and transfusions
   3. Absolute neutrophil count (ANC) ≥ 1000/mm^3 within 7 days before first dose of study treatment
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN) and total bilirubin ≤ 2.0 x ULN N (total bilirubin must be < 3 x ULN for patients with Gilbert's syndrome)

Exclusion Criteria:

1. Participant has any of the following conditions:

   1. Non secretory MM (Serum free light chains < 10 mg/dL)
   2. Solitary plasmacytoma
   3. Active plasma cell leukemia (ie, either 20% of peripheral white blood cells or > 2.0 x 109/L circulating plasma cells by standard differential)
   4. Waldenström macroglobulinemia (WM)
   5. Amyloidosis.
   6. Polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, skin changes (POEMS) syndrome
   7. Chronic respiratory disease that requires continuous oxygen
2. Significant cardiovascular disease, including but not limited to:

   1. Myocardial infarction ≤ 6 months before screening
   2. Ejection fraction ≤ 50%
   3. Unstable angina≤ 3 months before screening
   4. New York Heart Association Class III or IV congestive heart failure
   5. History of clinically significant arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
   6. Heart rate-corrected QT interval > 480 milliseconds based on Fridericia's formula
   7. History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place
   8. Uncontrolled hypertension at screening, defined as systolic blood pressure > 170 mmHg and diastolic blood pressure > 105 mmHg by ≥ 2 consecutive measurements. Prior therapy with sonrotoclax or other agents inhibiting BCL2 activity (eg, venetoclax)
3. Known infection with human immunodeficiency virus (HIV)
4. Serologic status reflecting active viral hepatitis B (HBV) or viral hepatitis C (HCV) infection as follows:

   1. Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Participants with presence of HBcAb, but absence of HBsAg, are eligible if HBV DNA is undetectable (limitation of sensitivity < 20 IU/mL) ,), and if they are willing to undergo monthly monitoring for HBV reactivation.
   2. Presence of HCV antibody. Participants with presence of HCV antibody are eligible if HCV RNA is undetectable (limitation of sensitivity < 15 IU/mL).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number Of Participants Experiencing Dose-limiting Toxicities (DLTs) | Up to 28 days
  DLTs will be based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 and will include most grade 3 or higher events, as defined in the protocol.
Part 1 And 2: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Adverse Events Leading to Discontinuation and Adverse Events of Special Interest (AESIs). | Up to 30 days after last dose of study drug
Part 2: Overall response rate (ORR) as Assessed by Investigator | Approximately 4 years
  Defined as the percentage of participants who achieved a stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) per International Myeloma Working Group (IMWG) criteria
Part 2: Very Good Partial Response (VGPR) or Better Response Rate as Assessed by Investigator | Upon study termination (Baseline up to first documentation of disease progression [PD] or death from any cause [approximately 4 years]
  Defined as the percentage of participants with a documented VGPR or better (including sCR, CR, and VGPR)
Part 2: Complete Response (CR) or Stringent Complete Response (sCR) as Assessed by Investigator | Upon study termination (Baseline up to first documentation of disease progression [PD] or death from any cause [approximately 4 years])
  defined as the percentage of participants with a documented CR or sCR

SECONDARY OUTCOMES:
Part 1: Area under the plasma concentration-time curve time 0 to the last measurable concentration (AUClast) After a Single Dose of Sonrotoclax | Cycle 1 (each cycle is up to 28 days)
Part 1: Maximum observed plasma concentration (Cmax) After a Single Dose of Sonrotoclax | Cycle 1 (each cycle is up to 28 days)
Part 1: Time to reach Cmax (tmax) After a Single Dose of Sonrotoclax | Cycle 1 (each cycle is up to 28 days)
Part 1: At Steady-state: AUC last, ss | Cycle 2 (each cycle is up to 28 days)
Part 1: At Steady-state: Cmax, ss | Cycle 2 (each cycle is up to 28 days)
Part 1: At Steady-state: trough plasma concentration (Ctrough) ss | Cycle 2 (each cycle is up to 28 days)
Part 1: At Steady-state: time to reach Cmax (tmax,ss) | Cycle 2 (each cycle is up to 28 days)
Part 2: Time to response (TTR) as Assessed by Investigator | Approximately 4 years
  TTR is defined as the time from start of treatment (for nonrandomized cohorts) or date of randomization (for randomized cohorts to first documentation of response of Partial Response (PR) or better
Part 2: Duration of response (DOR) as Assessed by Investigator | Approximately 4 years
  DOR is defined as the time from the date of the first documented response (PR or better) after treatment initiation until the date of first documented disease progression or death due to any cause, whichever occurs first. DOR will be analyzed only for patients who have achieved an overall response of at least PR. The distribution of DOR will be summarized by the Kaplan-Meier method.
Part 2: Progression-free survival (PFS) as Assessed by Investigator | Approximately 4 years
  PFS is defined as time from start of treatment （for nonrandomized cohorts） or date of randomization （for randomized cohorts） to the first documentation of disease progression or death, whichever occurs first
Part 2: Overall survival (OS) as Assessed by Investigator | Approximately 4 years
  OS defined as the time from start of treatment (for nonrandomized cohorts) or date of randomization (for randomized cohorts to the date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (84):
- United States (18):
  - University of Alabama At Birmingham Hospital, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - City of Hope At Irvine Lennar, Irvine, California
  - University of California At San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Emory University Winship Cancer Center, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College Newyork Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center Mskcc, New York, New York
  - The James Cancer Hospital and Solove Research Institute At Ohio State University, Columbus, Ohio
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Nepean Hospital, Kingswood, New South Wales
  - Monash Health, Clayton, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Brazil (7):
  - Hospital Sirio Libanes Brasilia, Brasília
  - Instituto Dor de Pesquisa E Ensino Distrito Federal, Brasília
  - Centro Gaucho Integrado de Oncologia Hospital Mae de Deus, Porto Alegre
  - Hospital Sao Rafael (Rede Dor), Salvador
  - Hospital Sirio Libanes, São Paulo
  - Instituto Dor de Pesquisa E Ensino Sao Paulo, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency the Vancouver Centre, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
- China (23):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Chao Yang Hospital, Beijing, Beijing Municipality
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital,the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Xianghu, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Fourth Peoples Hospital Affiliated to Tongji University, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciencestuanbo Branch, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Germany (4):
  - Universitaetsklinikum Aachen, Aachen
  - Universitatsklinikum Carl Gustav Carus An Der Technischen Universitat Dresden, Dresden
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Universitatsklinikum Wurzburg, Würzburg
- Greece (2):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - General Hospital of Athens Alexandra, Athens
- Sourasky Medical Center, Tel Aviv, Israel
- Italy (6):
  - Azienda Ospedaliera Policlinico Di Bari, Bari
  - Policlinico Sorsola Malpighi, Aou Di Bologna, Bologna
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori Irst, Meldola
  - Istituto Europeo Di Oncologia, Milan
  - Istituto Di Candiolo Irccs, Torino
  - Azienda Ospedaliera Universitaria Delle Marche, Torrette
- National University Hospital Singapore, Singapore, Singapore
- South Korea (5):
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, SeochoGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi
- Spain (4):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital Universitario Virgen Del Rocio, Seville
- United Kingdom (4):
  - Churchill Hospital Oxford University Hospital Nhs Trust, Headington
  - University College Hospital, London
  - Royal Marsden Nhs Foundation Royal Marsden Hospital, Sutton
  - Royal Cornwall Hospitalsnhs Trust, Truro

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/